CLINICAL TRIAL: NCT05058872
Title: Contraceptive Hormone and Reward Measurement (CHARM Study)
Acronym: CHARM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-3530
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Oral Hormonal Contraceptive Use; Neural Activity; Mood; Hedonic Function
Keywords: oral contraceptives; mood; reward processing; hedonic function
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levonorgestrel/ethinyl estradiol (Experimental): Levonorgestrel 0.15mg/ethinyl estradiol 0.03mg - once a day for 21 days
  Interventions: Drug: Levonorgestrel/ethinyl estradiol
- Placebo (Placebo Comparator): Placebo once a day for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levonorgestrel/ethinyl estradiol — Levonorgestrel 0.15mg/ethinyl estradiol 0.03mg
  Arms: Levonorgestrel/ethinyl estradiol
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
Purpose of this study: The purpose of this study is to learn more about how hormonal oral contraceptives affect brain processes and emotional wellbeing.

Procedures: If participants agree to participate, the following will happen:

1. Eligibility visit (remote screening session)
2. If participants are eligible to participate in the study, they will be placed in one of two groups. If they are in the first group, they will be asked to take an oral contraception pill ("study drug") every day for 21 days. If they are in the second, they will take a placebo every day for 21 days. A placebo is a pill that looks like medicine but is not real and will have no medical effect on participants. Participants will not get to choose which group they are in, nor will they be told which group they are in.
3. During the three-week period in which participants will take either the study drug or placebo, they will be asked to complete daily check-in surveys on their computer or mobile device.
4. Participants will be asked to attend two additional visits over the course of about three weeks. At these visits, participants will be asked to undergo a urine drug screen, a blood draw, and a magnetic resonance imaging (MRI). They will also be asked to complete behavioral questionnaires.

DETAILED DESCRIPTION:
Hypothesis:

The principal investigator hypothesizes that treatment with oral contraceptives, specifically a combination of a synthetic estrogen and progestin, in adult females will result in deficits in reward processing.

Specific Aims:

1. Subjective ratings of mood and hedonic function. Based on previous evidence, the principal investigator hypothesizes that H1a) treatment with a hormonal oral contraceptive will result in decreased self-reports of sexual function and interest/enjoyment in non-sexual pleasurable activities as measured by the Sexual Function Questionnaire and Dimensional Anhedonia Rating Scale, respectively.
2. Neural activity in reward processing areas during an incentive delay task. Via functional magnetic resonance imaging, neural activity will be measured during both the anticipation and receipt of a pleasurable image (erotica, pleasant images of the outdoors, and "cute" animals). Activation of nucleus accumbens and ventromedial pre-frontal cortex is positively associated with feelings of anticipation and pleasure, respectively (10). The principal investigator hypothesizes that H2) treatment with a hormonal oral contraceptive will result in decreased activity in these regions, consistent with decreased reward anticipation and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and older;
2. Right-handed;
3. Assigned female at birth;
4. Regular 21-35 day menstrual cycles for the past 6 months per self-report;
5. In generally good health per self-report. Those with a chronic medical condition may participate at the discretion of the principal investigator if the condition is stable;
6. Willingness to abstain from intercourse or use a non-hormonal back-up method of contraception (e.g., condoms) during the entire course of the study;
7. Negative urine drug screen, excepting marijuana or benzodiazepine that is being prescribed by a physician as a sleep aid, assessed at the baseline visit;
8. Ability to abstain from caffeine and/or cannabis for 2 hours prior to functional Magnetic Resonance Imaging (fMRI) scan visits;
9. Access to a reliable internet connection or cell phone data to complete daily questionnaires;
10. For those wishing to complete study screening session remotely: access to a reliable internet connection, computer to complete electronic consent and a private space to complete the session.

Exclusion Criteria:

1. Presence or history of severe or unstable physical, neurological (per health history interview) or psychiatric disorders (assessed by Miniature International Neuropsychiatric Interview (MINI) but per Diagnostic and Statistical Manual of Mental Disorders - fifth edition (DSM-V) criteria, and the discretion of the principal investigator);
2. Lifetime history of psychotic disorders;
3. History of substance use disorder that has not been in remission (as defined by a substance free period of at least one year). However, individuals with mild disorders, disorders solely limited to cannabis, and/or those who have achieved close to one year of remission may be eligible at the discretion of the PI;
4. Presence or history of any category 3 or 4 conditions or medications per the CDC's (Centers for Disease Control and Prevention) Medical Eligibility Criteria for Contraceptive Use pertaining to combined hormonal contraceptive methods as per self-report and reviewed by the principal investigator;
5. Irregular menstrual periods per self-report;
6. Any current tobacco smoking (former smokers are eligible so long as their quit date was greater than one year ago);
7. Any personal or family history of a venous thromboembolism;
8. Known diagnosis of hypertensive disorder;
9. Any current or past history of malignancy;
10. Migraines with aura;
11. Systolic blood pressure greater than or equal to 140 or diastolic pressure greater than or equal to 90 taken at baseline visit;
12. Currently nursing an infant;
13. Known chromosomal or hormonal disorder affecting sex steroids;
14. Use of hormonal contraceptives currently or in the past 3 months, or use of medications that directly affect sex hormones (i.e. gonadotropin releasing hormone agonists, selective estrogen receptor modifiers);
15. Current pregnancy or pregnancy/delivery in the past six months;
16. Intention to become pregnant during study participation;
17. Current use of psychotropic medication;
18. Claustrophobia;
19. Metal in body unsafe for magnetic resonance imaging;
20. Weight over 300 pounds;
21. Conditions that would make magnetic resonance imaging unsafe for participants (i.e. aneurysm clip, cardiac pacemaker, etc.).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in ratings of anhedonia after 21 days of receiving either levonorgestrel/ethinyl estradiol or placebo as measured by the Dimensional Anhedonia Rating Scale | Baseline, 21 days post-intervention
  The Dimensional Anhedonia Rating Scale is validated measure of anhedonia (lack of pleasure, desire, and motivation). Scores range from 17 to 85 with higher scores reflecting a better outcome/less anhedonia
Change in ratings of sexual function after 21 days of receiving either levonorgestrel/ethinyl estradiol or placebo as measured by the Female Sexual Function Index. | Baseline, 21 days post-intervention
  The Female Sexual Function Index is a validated questionnaire of various domains of sexual functioning in women. Scores range from 2 to 36, with higher scores reflecting better outcomes/better sexual function.
Change in Blood Oxygen Level Dependent (BOLD) Signal after 21 days of treatment with either levonorgestrel/ethinyl estradiol or placebo | Baseline, 21 days post-intervention
  Blood-oxygen-level dependent contrast imaging, or BOLD-contrast imaging, is a method used in functional magnetic resonance imaging (fMRI) to observe different areas of the brain or other organs, which are found to be active at any given time. BOLD signal in the brain will be measured during a reward task both at baseline and after 21 days of receiving either levonorgestrel/ethinyl estradiol or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Novick, MD PhD, Principal Investigator — University of Colorado Denver Anschutz Medical Campus
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No